CLINICAL TRIAL: NCT02044367
Title: Relative Bioavailability of Dabigatran After Administration of Different Dosage Forms of Multiple Doses of 150 mg Dabigatran Etexilate (Hard Capsule, Granules Resolved in Reconstitution Solution, Pellets on Food) in Healthy Male Volunteers (an Open-label, Randomised, Multiple-dose, Three Way Crossover Study)
Brief Title: Relative Bioavailability of Dabigatran Capsules, Pellets and Oral Solution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.194; 2013-002498-23 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

ARMS (3):
- Test 1 (Treatment A) (Experimental): multiple dose of dabigatran
  Interventions: Drug: Dabigatran etexilate
- Test 2 (Treatment B) (Experimental): multiple dose of dabigatran
  Interventions: Drug: Dabigatran etexilate
- Reference (Experimental): multiple dose of dabigatran
  Interventions: Drug: Dabigatran etexilate

INTERVENTIONS:
Drug: Dabigatran etexilate — Pellets (multiple dose of dabigatran)
  Arms: Test 1 (Treatment A)
Drug: Dabigatran etexilate — Granules resolved in reconstitution solution (multiple dose of dabigatran)
  Arms: Test 2 (Treatment B)
Drug: Dabigatran etexilate — Hard capsule (multiple dose of dabigatran)
  Arms: Reference

SUMMARY:
To investigate the relative bioavailability of dabigatran etexilate as pellets on food and of dabigatran etexilate as granules resolved in reconstitution solution, each with dabigatran etexilate as capsule following oral administration. To evaluate acceptability and palatability of Pellets sprinkled on food and Oral Liquid Formulation

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to the investigator's assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (Blood Pressure, Pulse Rate), 12-lead electrocardiogram, and clinical laboratory tests
2. Age 18 to 55 years (incl.)
3. Body Mass Index 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

1. Any finding in the medical examination (including Blood Pressure, Pulse Rate or electrocardiogram) deviating from normal and judged clinically relevant by the investigator.
2. Repeated measurement of systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug
7. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders
8. Subjects who in the investigator's judgement are perceived as having an increased risk of bleeding, for example because of:

   * Hemorrhagic disorders or bleeding diathesis
   * Occult blood in faeces or haematuria
   * Trauma or surgery within the last month or as long as an excessive risk of bleeding persists after these events, or planned surgery during trial participation
   * History of arteriovenous malformation or aneurysm
   * History of gastroduodenal ulcer disease or gastrointestinal haemorrhage
   * History of intracranial, intraocular, spinal, retroperitoneal, or atraumatic intraarticular bleeding
   * Anemia at screening
   * Thrombocytopenia (platelet count less than 100/nL)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1160.194.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- T1-T2-R: T1: pellets on food; T2: granules for reconstitution into solution; R: hard capsule. The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for all treatments T1, T2 and R. All treatments were administered orally with 240 mL of water.
- T1-R-T2: T1: pellets on food; R: hard capsule; T2: granules for reconstitution into solution. The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for all treatments T1, T2 and R. All treatments were administered orally with 240 mL of water.
- T2-T1-R: T2: granules for reconstitution into solution; T1: pellets on food; R: hard capsule. The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for all treatments T1, T2 and R. All treatments were administered orally with 240 mL of water.
- T2-R-T1: T2: granules for reconstitution into solution; R: hard capsule; T1: pellets on food. The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for all treatments T1, T2 and R. All treatments were administered orally with 240 mL of water.
- R-T1-T2: R: hard capsule; T1: pellets on food; T2: granules for reconstitution into solution. The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for all treatments T1, T2 and R. All treatments were administered orally with 240 mL of water.
- R-T2-T1: R: hard capsule; T2: granules for reconstitution into solution; T1: pellets on food. The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for all treatments T1, T2 and R. All treatments were administered orally with 240 mL of water.
Period: Overall Study
Arm/Group | T1-T2-R | T1-R-T2 | T2-T1-R | T2-R-T1 | R-T1-T2 | R-T2-T1
Started | 9 | 9 | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The evaluation of demographic and baseline characteristics were performed on the treated set which included all subjects who received at least 1 dose of study drug.
Groups:
- Overall: A randomised, open-label, 3-way crossover, multiple dose trial consisting of 3 identical treatment periods of 3 days. Study drug (150 mg dabigatran etexilate) was administrated twice daily on Day 1 and Day 2 and once on Day 3. The dosage forms used were: hard capsule, granules resolved in reconstitution solution and pellets on food. Treatment periods were separated by a washout phase of at least 5 days between last drug administration of one treatment and the first drug administration of the next treatment.
Arm/Group | Overall
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval t for Total Dabigatran.
Description: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t for total dabigatran.
Time Frame: 47:55, 48:30, 49:00, 49:30, 50:00, 50:30, 51:00, 51:30, 52:00, 54:00, 56:00, 58:00, 60:00 relative to first drug administration
Population: Pharmacokinetic analysis set (PKS) included all treated subjects that provided at least 1 observation for at least 1 primary or secondary PK endpoint without relevant protocol deviations with respect to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng∙h/mL
Groups:
- T1 (Treatment A): multiple dose of dabigatran (Pellets)
  The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for all treatments T1, T2 and R. All treatments were administered orally with 240 mL of water.
- T2 (Treatment B): multiple dose of dabigatran (Granules resolved in reconstitution solution)
  The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for all treatments T1, T2 and R. All treatments were administered orally with 240 mL of water.
- R (Reference): multiple dose of dabigatran (Hard capsule)
  The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for all treatments T1, T2 and R. All treatments were administered orally with 240 mL of water.
Arm/Group | T1 (Treatment A) | T2 (Treatment B) | R (Reference)
Number analyzed (Participants) | 54 | 54 | 53
ng∙h/mL | 1220 (34.1) | 1160 (27.0) | 893 (46.8)
Statistical Analysis 1: Comparison: T1 (Treatment A) vs R (Reference); Analysis of variance (ANOVA) on the logarithmic scale was used including effects for 'sequence', 'period' and 'treatment' as fixed effects and 'subjects within sequences' as random effect. CIs were calculated based on the residual error from ANOVA; Test type: Non-Inferiority or Equivalence — The sample size determination was not based on a power calculation, but to assure a precise estimation of the relative bioavailability. For this 3-way crossover trial, a precision (defined by ratio of upper CI limit to adjusted GMR) of at most 1.17 had been considered necessary and sufficient by the project team; gMean Ratio T1/R (%) = 137.01, 90% CI 2-sided [125.773 to 149.250], Standard Deviation 26.8 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: T2 (Treatment B) vs R (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean Ratio T2/R (%) = 130.43, 90% CI 2-sided [119.628 to 142.200], Standard Deviation 27.1 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV)

2. Primary Outcome: Maximum Measured Concentration of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval t for Total Dabigatran.
Description: Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t for total dabigatran.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | T1 (Treatment A) | T2 (Treatment B) | R (Reference)
Number analyzed (Participants) | 54 | 54 | 53
ng/mL | 191 (37.4) | 184 (27.3) | 131 (50.8)
Statistical Analysis 1: Comparison: T1 (Treatment A) vs R (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean Ratio T1/R (%) = 146.16, 90% CI 2-sided [132.217 to 161.576], Standard Deviation 31.6 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: T2 (Treatment B) vs R (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean Ratio T2/R (%) = 141.06, 90% CI 2-sided [127.644 to 155.876], Standard Deviation 31.5 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV)

3. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval t for Free Dabigatran.
Description: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t for free dabigatran.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | T1 (Treatment A) | T2 (Treatment B) | R (Reference)
Number analyzed (Participants) | 54 | 54 | 53
ng*h/mL | 1000 (35.8) | 958 (27.6) | 727 (50.8)
Statistical Analysis 1: Comparison: T1 (Treatment A) vs R (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean Ratio T1/R (%) = 137.61, 90% CI 2-sided [126.418 to 149.797], Standard Deviation 26.5 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: T2 (Treatment B) vs R (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean Ratio T2/R (%) = 132.00, 90% CI 2-sided [120.714 to 144.342], Standard Deviation 28.0 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV)

4. Secondary Outcome: Maximum Measured Concentration of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval t for Free Dabigatran.
Description: Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t for free dabigatran.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | T1 (Treatment A) | T2 (Treatment B) | R (Reference)
Number analyzed (Participants) | 54 | 54 | 53
ng/mL | 157 (37.9) | 154 (27.6) | 106 (55.1)
Statistical Analysis 1: Comparison: T1 (Treatment A) vs R (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean Ratio T1/R (%) = 147.80, 90% CI 2-sided [133.384 to 163.779], Standard Deviation 32.4 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: T2 (Treatment B) vs R (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean Ratio T2/R (%) = 144.80, 90% CI 2-sided [130.853 to 160.242], Standard Deviation 32.0 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV)

5. Secondary Outcome: Acceptability Rating for Pellets (on Food) and Oral Solution Will be Assessed by Asking the Subjects 1 Multiple Choice Verbal Question.
Description: Acceptability question: "Would you accept to take this medication for chronic use?" with 3 possible answers: Yes - No - I am not sure.
Time Frame: once on day 3 (48 hours after first dose)
Population: Treated set including all subjects that provided at least 1 observation for at least 1 of the questions for at least 1 of the test products.
Measure: Number; unit: participants
Groups:
- T1 (Treatment A): T1: Pellets on food The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for both treatments T1 and T2. All treatments were administered orally with 240 mL of water.
- T2 (Treatment B): T2: Granules resolved in reconstitution solution The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for both treatments T1 and T2. All treatments were administered orally with 240 mL of water.
Arm/Group | T1 (Treatment A) | T2 (Treatment B)
Number analyzed (Participants) | 53 | 53
participants
  Yes | 37 | 29
  No | 9 | 17
  I am not sure | 7 | 7

6. Secondary Outcome: Palatability Rating for Pellets (on Food) and Oral Solution Will be Assessed by Asking the Subjects 1 Multiple Choice Verbal Question.
Description: Palatability question: "How do you rank the taste?" with 5 possible answers: Very good - Good - Fair - Acceptable - Not acceptable.
Time Frame: once on day 3 (48 hours after first dose)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | T1 (Treatment A) | T2 (Treatment B)
Number analyzed (Participants) | 53 | 53
participants
  Very good | 2 | 0
  Good | 20 | 15
  Fair | 18 | 17
  Acceptable | 11 | 14
  Not acceptable | 2 | 7

ADVERSE EVENTS:
Time Frame: First dose of study drug date/time until the end-of-trial examination (last per protocol visit)
Groups:
- T1 (Treatment A): multiple dose of dabigatran (Pellets). The treatments were 150 mg dabigatran etexilate twice daily on Days 1 and 2 and once after an overnight fast of at least 10 hours on Day 3 for all treatments T1, T2 and R. All treatments were administered orally with 240 mL of water.
Arm/Group | T1 (Treatment A) | T2 (Treatment B) | R (Reference)
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 2/54 | 3/54 | 1/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T1 (Treatment A) (N=54) | T2 (Treatment B) (N=54) | R (Reference) (N=54)
Headache (Nervous system disorders) | 2 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes